CLINICAL TRIAL: NCT02119780
Title: Clinical Study to Evaluate the Efficacy and Safety of YVOIRE® Contour Compared With Restylane SubQ™ Injected Into the Anteromedial Malar Region
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LG-HACL014
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Normal, Healthy Adults With Moderate, Severe, or Very Severe Volume Loss of Anteromedial Malar Region

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- YVOIRE® contour (Experimental)
  Interventions: Device: YVOIRE® contour
- Restylane SubQ™ (Active Comparator)
  Interventions: Device: Restylane SubQ™

INTERVENTIONS:
Device: YVOIRE® contour — YVOIRE® contour injection into the anteromedial malar region
  Arms: YVOIRE® contour
Device: Restylane SubQ™ — Restylane SubQ™ injection into the anteromedial malar region
  Arms: Restylane SubQ™

SUMMARY:
This study is purposed to evaluate the efficacy and safety of YVOIRE® contour compared with Restylane SubQ™ injected into the anteromedial malar region.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, 20-65 years of age
* Have anteromedial malar region volume loss as grade 2, 3, or 4 on the Mid Face Aesthetic Scale (MFAS) symmetrically on both sides
* Desire filler treatment to correct volume loss in the anteromedial malar region
* Accept the obligation not to receive any other mid facial procedures or treatments during the study
* Signed informed consent
* Those who fall under one of the following 3 cases

  1. Males or females who are surgically sterile
  2. Post-menopausal females who are above 45 years of age and 2 years after the last menstruation
  3. Fertile premenopausal females or males without having a surgical sterilization, who have agreed to use at least two contraception methods (one of the barrier methods must be included) for up to 14 days after the last treatment of the investigational device to avoid pregnancy

Exclusion Criteria:

* Have a history of hypertrophic scars or keloids
* Other criteria as identified in the protocol

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Mid Face Aesthetic Scale (MFAS) score | 26 weeks after treatment
  Mean of MFAS score as assessed by the independent blinded rater

SECONDARY OUTCOMES:
Mid Face Aesthetic Scale (MFAS) score | 2, 14, and 52 weeks after treatment
  Mean of MFAS score as assessed by the independent blinded rater
Mid Face Aesthetic Scale (MFAS) score | 2, 14, 26, and 52 weeks after treatment
  Changes of MFAS score as assessed by the independent blinded rater
Mid Face Aesthetic Scale (MFAS) Responder rate | 2, 14, 26, and 52 weeks after treatment
  MFAS Responder (at least a one-point improvement on the MFAS) rate as assessed by the independent blinded rater
Global Aesthetic Improvement Scale (GAIS) score | 2, 14, 26, and 52 weeks after treatment
  Mean of GAIS score as assessed by subject
Global Aesthetic Improvement Scale (GAIS) Responder rate | 2, 14, 26, and 52 weeks after treatment
  GAIS Responder (at least a one-point improvement on the GAIS) rate as assessed by subject

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea